CLINICAL TRIAL: NCT03437967
Title: Effect of LASER Photobiomodulation Therapy on Chronic Pain and Opioid Weaning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient withdrawal symptoms unblinded the study
Sponsor: LiteCure LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBMT for Chronic Pain
Record Dates: First submitted 2017-12-21; First posted 2018-02-19 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Low-Level Light Therapy; Laser Therapy

STUDY DESIGN:
Intervention Model Description: This is a prospective interventional study using a double-blind 4-period crossover design to assess the efficacy of LASER Photobiomodulation therapy compared to sham (LOW POWER LASER) therapy in reducing pain and improving compliance with OPM weaning. LASER photobiomodulation treatments or sham treatments will be provided three times a week using standardized protocols. Crossover will occur every 3 weeks with weekly data collection occurring at the end of each week allowing for washout and to minimize the carryover effects of active treatment. Data collection will consist of LASER and sham treatments, prescribed pain medication dosage and quantity, subjective pain questionnaires, and urine samples. Cognitive and memory screening will occur every 3 weeks at the end of each period prior to crossover.
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham therapy will consist of treatment using an identically appearing device that delivers low level LASER POWER to simulate LASER treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ABAB (Other): Treatment, either LASER (arm A) or LOW LEVEL LASER (arm B) will be provided 3 (not less than 2) days a week for three weeks at which time crossover into the alternate arm occurs (BABA to ABAB or ABAB to BABA).
  ABAB initial period is active treatment - LASER.
  Active Treatment:
  LASER light is delivered to the skin and deeper tissues affected by pain using either a wand or glass roller ball. Ten to 25 Watts of LASER energy is delivered to the painful regions for 8 to 16 minutes depending on the size of the area treated and other factors such as skin pigmentation.
  Interventions: Device: LightForce EXPi
- BABA (Other): Treatment, either LASER (arm A) or LOW LEVEL LASER (arm B) will be provided 3 (not less than 2) days a week for three weeks at which time crossover into the alternate arm occurs (BABA to ABAB or ABAB to BABA).
  BABA initial period is sham treatment - LOW LEVEL LASER.
  LOW LEVEL LASER "treatment":
  Low level LASER is provided in a similar fashion using LASER power levels (1 Watt) that produce warmth only at superficial skin levels.
  Interventions: Device: LightForce EXPi

INTERVENTIONS:
Device: LightForce EXPi — LASER photobiomodulation therapy of 15-25 watts of coherent infrared light to affected area for 10 minutes using wand-type probe.
  Other Names: LASER photobiomodulation therapy; LASER therapy

SUMMARY:
This study will examine the effect of LASER photobiomodulation therapy on pain and opioid pain medication weaning on patients who are undergoing opioid pain medication weaning.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if treatment with LASER photobiomodulation therapy reduces pain and facilitates opioid pain medication (OPM) reduction (weaning). The subject group includes patients with chronic pain who are undergoing OPM weaning and are candidates for LASER photobiomodulation therapy. This is a prospective interventional study using a double-blind 4-period crossover design to assess the efficacy of HIGH POWER LASER photobiomodulation therapy compared to sham (LOW POWER LASER) therapy in reducing pain and improving compliance with OPM weaning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Taking prescribed opioid pain medications in an amount in excess of 30 Morphine Equivalent Dose (MED) for 6 months or longer.
* Have been recommended to wean or reduce their MED.
* Medically stable such that subject does not have unstable angina, COPD requiring supplemental oxygen, untreated or active cancer or similar conditions that would make participation difficult or unsafe.
* Compliant with all physician recommendations relating to medication usage.
* Ambulatory and able to use the toilet independently.
* Negative pregnancy test in subjects of childbearing potential
* Willing to attempt opioid pain medication taper.
* Competent to provide informed consent.
* Capable of understanding and completing study questionnaires.
* Subject willing to participate in the study for up to 12 weeks.

Exclusion Criteria:

* Not capable of understanding or completing study questionnaires.
* Lacking capacity to provide fully informed consent.
* Substance use disorder not in remission.
* Considering surgery or other invasive procedures that would take place during the study.
* Used isotretinoin (Accutane) within 6 months prior to study enrollment
* Cancer not in remission.
* Need of ongoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy, massage therapy, chiropractic care or other treatments intended to remediate pain other than treatment in the Sharp Pain Program.
* A female who is pregnant or lactating, or of childbearing potential unless a medically acceptable method of birth control is in use.
* Any use of light-activated drugs (photodynamic therapy) or heat sensitive medications within 30 days of first treatment.
* Used an investigational drug/device therapy or participated in any clinical investigation relating to pain within 4 weeks prior to study enrollment.
* A psychiatric or psychological condition that would place undo stress on the subject, prevent full participation or compromise data collection.
* The subject is otherwise determined, based on the opinion of the Investigator, to be an unsuitable candidate for enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Compliance with Medical Opioid Use Reduction Protocol | 12 weeks
  Prescriptions for pain medications will be provided each week. Each successive prescription will have a decreasing quantity of tablets consistent with an agreed upon taper rate. Taper rates will be roughly based upon the recommendations of the CDC (10% per week). Subjects will have the option of postponing the taper by one week as often as every other week. If a subject was to exercise every option available to them to delay taper, then the weaning process would take twice as long and the rate of taper would be cut in half.
  The study will compare the number of missed medication tapers, and the taper rates of patients in the HIGH POWER LASER treatment periods to those in the LOW LEVEL LASER THERAPY treatment periods.

SECONDARY OUTCOMES:
Self-reported measure of Pain. | 12 weeks
  Participants will complete the Visual Analogue Scale for Pain (Wong Baker FACES pain rating scale), taken at baseline, weekly thereafter, and immediately after the last treatment.
Self-reported measure of Quality of Life. | 12 weeks
  Participants will complete the 36-Item Short Form Health Survey (SF36) at baseline and at study completion.
Self-reported measure of Depression. | 12 weeks
  Participants will complete the 17-item Hamilton Depression Rating Scale (HAM-D) at baseline and at study completion.
Self-reported measure of Anxiety. | 12 weeks
  Participants will complete the 40-item State-Trait Anxiety Inventory (STAI) at baseline and at study completion.
Self-reported measure of Sleep Quality. | 12 weeks
  Participants will complete the Pittsburgh Sleep Quality Index (PSQI) at baseline and at study completion.
Urine screening | 12 weeks
  Weekly urine screening will be conducted to assess deviations from treatment (use of non prescribed medications or substances).

CONTACTS AND LOCATIONS:
Overall Officials: Jerome C Stenehjem, Md, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Alison DeRose Rehabilitation Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no intent to share data and no plan formulated at this time.